CLINICAL TRIAL: NCT00979901
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Study Investigating the Clinical Effects of Montelukast in Patients With Seasonal Allergic Rhinitis--Spring Study
Brief Title: Montelukast in Patients With Seasonal Allergic Rhinitis - Spring 2000 Study (MK-0476A-162)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476A-162; MK0476A-162; 2009_664
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2010-06-08 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Loratadine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): montelukast
  Interventions: Drug: Comparator: montelukast
- 2 (Experimental): loratadine
  Interventions: Drug: Comparator: loratadine
- 3 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: placebo
- 4 (Experimental): montelukast/loratadine
  Interventions: Drug: Comparator: montelukast/loratadine

INTERVENTIONS:
Drug: Comparator: montelukast — 10 mg montelukast tablet given once daily at bedtime for 2 weeks
  Arms: 1
Drug: Comparator: loratadine — 10 mg loratadine tablet given once daily at bedtime for 2 weeks
  Arms: 2
Drug: Comparator: placebo — placebo tablet given once daily at bedtime for 2 weeks
  Arms: 3
Drug: Comparator: montelukast/loratadine — montelukast 10-mg/loratadine 10-mg combination tablet taken orally once daily at bedtime for 2 weeks
  Arms: 4

SUMMARY:
This study will evaluate the ability of montelukast to improve the signs and symptoms of seasonal allergic rhinitis compared with loratadine and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a documented history of seasonal allergic rhinitis symptoms that flare up during the study season
* Patient is a nonsmoker and has been a nonsmoker for at least 1 year
* Patient is in good general health

Exclusion Criteria:

* Patient is hospitalized
* Patient is a woman who is less than 8 weeks postpartum or is breast-feeding
* Patient intends to move or vacation away during the study
* Patient has had any major surgery within 4 weeks of study start
* Patient is a current or past abuser of alcohol or illicit drugs
* Patient has been treated in an emergency room for asthma in the past month
* Patient had an upper respiratory infection with in 3 weeks prior to study start

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1577 (Actual)
Dates: Start 2000-03; Primary Completion 2000-05 (Actual); Study Completion 2000-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Philip G, Malmstrom K, Hampel FC, Weinstein SF, LaForce CF, Ratner PH, Malice MP, Reiss TF; Montelukast Spring Rhinitis Study Group. Montelukast for treating seasonal allergic rhinitis: a randomized, double-blind, placebo-controlled trial performed in the spring. Clin Exp Allergy. 2002 Jul;32(7):1020-8. doi: 10.1046/j.1365-2222.2002.01422.x. PMID 12100048

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 50 sites (43 in the US and 7 in Canada).
  Primary Therapy Period: March 2000 to July 2000.
Pre-assignment Details: Patients who required excluded medication and those who did not meet a minimum predefined level of combined daytime nasal symptoms score during the run-in period were excluded from randomization.
Groups:
- Placebo: Matching-image placebo tablet to each of montelukast, loratadine, and montelukast/loratadine combination taken orally once daily at bedtime for 2 weeks.
- Montelukast 10 mg: Montelukast 10 mg tablet, loratadine matching-image placebo tablet, and montelukast/loratadine matching-image placebo tablet taken orally once daily at bedtime for 2 weeks.
- Loratadine 10 mg: Montelukast matching-image placebo tablet, loratadine 10 mg tablet, and montelukast/loratadine matching-image placebo tablet taken orally once daily at bedtime for 2 weeks.
- Montelukast/Loratadine: Montelukast matching-image placebo tablet, loratadine matching-image placebo tablet, and montelukast 10 mg/loratadine 10 mg combination tablet taken orally once daily at bedtime for 2 weeks. During the study, patients in the montelukast/loratadine combination treatment group were discontinued from further participation due to a business decision by the sponsor.
Period: Overall Study
Arm/Group | Placebo | Montelukast 10 mg | Loratadine 10 mg | Montelukast/Loratadine
Started | 352 | 348 | 602 | 275
Completed | 334 | 336 | 573 | 159
Not Completed | 18 | 12 | 29 | 116
Not completed — Adverse Event | 1 | 3 | 9 | 2
Not completed — Lack of Efficacy | 8 | 4 | 9 | 0
Not completed — Lost to Follow-up | 1 | 1 | 2 | 0
Not completed — Protocol Violation | 2 | 2 | 7 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 1
Not completed — Noncompliance | 1 | 0 | 0 | 0
Not completed — out-of-state | 1 | 0 | 0 | 0
Not completed — vacation | 1 | 0 | 0 | 0
Not completed — elevated lab values pre-randomization | 1 | 0 | 0 | 0
Not completed — Discontinued in Error | 0 | 1 | 0 | 0
Not completed — Left Country | 0 | 0 | 1 | 0
Not completed — Treatment Group Terminated by Sponsor | 0 | 0 | 0 | 112

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Montelukast 10 mg | Loratadine 10 mg | Montelukast/Loratadine | Total
Number analyzed (Participants) | 352 | 348 | 602 | 275 | 1577
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.9 (12.4) | 36.5 (12.6) | 36.3 (13.0) | 37.1 (11.95) | 36.39 (12.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 229 | 233 | 390 | 184 | 1036
  Male | 123 | 115 | 212 | 91 | 541
Daytime eye symptoms score [Mean (Standard Deviation); unit: Units on a Scale] — Computed using the average values of the 4 individual daytime eye symptoms scores of tearing, itching, red, and puffy eyes. Scores were measured as 0 (best) to 3 (worst). Baseline is computed as the average daily value during the run-in period.
  Units on a Scale | 1.44 (0.78) | 1.39 (0.77) | 1.40 (0.76) | 0 (0) | 1.41 (0.77)
Daytime nasal symptoms score [Mean (Standard Deviation); unit: Units on a Scale] — Computed using the average values of the 4 individual daytime nasal symptoms scores of congestion, rhinorrhea, itching, and sneezing. Scores were measured as 0 (best) to 3 (worst). Baseline is computed as the average daily value during the run-in period.
  Units on a Scale | 2.10 (0.43) | 2.09 (0.44) | 2.06 (0.41) | 0 (0) | 2.08 (0.43)
Nighttime symptoms score [Mean (Standard Deviation); unit: Units on a Scale] — Computed using the average values of the 3 individual nighttime symptoms scores of nasal congestion upon awakening, difficulty going to sleep, and nighttime awakenings. Scores were measured as 0 (best) to 3 (worst). Baseline is computed as the average daily value during the run-in period.
  Units on a Scale | 1.46 (0.66) | 1.43 (0.64) | 1.45 (0.64) | 0 (0) | 1.45 (0.65)
Rhinoconjunctivitis quality-of-life questionnaire (RQLQ) overall score [Mean (Standard Deviation); unit: Units on a Scale] — Computed by averaging the scores of the 7 domains of activity, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotions. Scores were measured as 0 (best) to 6 (worst). The 7 domains included 28 questions total. The average score was calculated for each domain, then the 7 domains were averaged to obtain the overall score. Baseline is the Visit 3 value.
  Units on a Scale | 3.22 (0.99) | 3.12 (0.99) | 3.09 (1.03) | 0 (0) | 3.13 (1.01)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Daytime Nasal Symptoms Score Over 2 Weeks
Description: Mean change from baseline in Daytime Nasal Symptoms score.
  Patients were asked to rate each of the 4 nasal symptoms of Congestion, Rhinorrhea, Itching, and Sneezing daily
  on a 4-point scale. The average of the 4 individual nasal symptoms scores was reported as the Daytime Nasal
  Symptoms Score. Scores were measured as 0 (best) to 3 (worst).
Time Frame: Baseline and Week 2
Population: The primary efficacy analysis was based on the ITT (all-patients treated) principle, i.e., all patients who had a baseline and at least one posttreatment measurement were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast 10 mg | Loratadine 10 mg
Number analyzed (Participants) | 351 | 344 | 599
Units on a Scale | -0.24 [-0.29 to -0.18] | -0.37 [-0.43 to -0.31] | -0.47 [-0.52 to -0.43]

2. Secondary Outcome: Mean Change From Baseline in Nighttime Symptoms Score Over 2 Weeks
Description: Mean change from baseline in Nighttime Symptoms Score.
  Patients were asked to rate each symptom daily on a 4-point scale, and the combined score of Nasal Congestion Upon Awakening, Difficulty Going to Sleep, and Nighttime Awakenings was reported as the Nighttime Symptoms Score. Scores were measured as 0 (best) to 3 (worst).
Time Frame: Baseline and Week 2
Population: The secondary efficacy analyses were based on the ITT (all-patients treated) principle, i.e., all patients who had a baseline and at least one posttreatment measurement were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast 10 mg | Loratadine 10 mg
Number analyzed (Participants) | 351 | 345 | 598
Units on a Scale | -0.14 [-0.19 to -0.09] | -0.27 [-0.32 to -0.22] | -0.23 [-0.27 to -0.19]

3. Secondary Outcome: Mean Change From Baseline in Daytime Eye Symptoms Score Over 2 Weeks
Description: Mean change from baseline in Daytime Eye Symptoms scores.
  Patients were asked to rate each of the 4 eye symptoms of tearing, itchy, red, and puffy eyes daily on a 4-point scale. The average of the 4 individual eye symptoms scores was reported as the Daytime Eye Symptoms Score. Scores were measured as 0 (best) to 3 (worst).
Time Frame: Baseline and Week 2
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast 10 mg | Loratadine 10 mg
Number analyzed (Participants) | 351 | 344 | 599
Units on a Scale | -0.12 [-0.17 to -0.06] | -0.26 [-0.32 to -0.20] | -0.32 [-0.36 to -0.28]

4. Secondary Outcome: Patient's Global Evaluation of Allergic Rhinitis at Week 2
Description: An evaluation by the patient, administered at the last visit (or
  upon discontinuation) using a 7-point scale, of the change in symptoms as compared to the beginning of the
  study. Scores were measured as 0 (best) to 6 (worst).
Time Frame: Week 2
Population: This secondary endpoint analysis was performed using the intention-to-treat approach. Patients were excluded if no treatment period data were available. No missing values were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast 10 mg | Loratadine 10 mg
Number analyzed (Participants) | 347 | 343 | 595
Units on a Scale | 2.62 [2.46 to 2.79] | 2.20 [2.04 to 2.36] | 2.13 [2.01 to 2.25]

5. Secondary Outcome: Physician's Global Evaluation of Allergic Rhinitis at Week 2
Description: An evaluation by the physician, administered at the last visit (or upon discontinuation) using a 7-point scale, of the change in symptoms as compared to the beginning of the study. Scores were measured as 0 (best) to 6 (worst).
Time Frame: Week 2
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast 10 mg | Loratadine 10 mg
Number analyzed (Participants) | 347 | 343 | 594
Units on a Scale | 2.53 [2.38 to 2.67] | 2.23 [2.08 to 2.37] | 2.17 [2.06 to 2.29]

6. Secondary Outcome: Mean Change From Baseline in Rhinoconjunctivitis Quality-of-life Questionnaire (RQLQ) Overall Score at Week 2
Description: Patients completed the validated, self-administered RQLQ, which included 28 items on a 7-point scale across 7 domains: activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional. Scores for each domain were averaged, then scores for the 7 domains were averaged for the overall score. Scores were measured as 0 (best) to 6 (worst).
Time Frame: Week 2
Population: This secondary endpoint analysis was performed using the intention-to-treat approach. Patients were excluded if no baseline or treatment period data were available. No missing values were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast 10 mg | Loratadine 10 mg
Number analyzed (Participants) | 348 | 344 | 598
Units on a Scale | -0.65 [-0.76 to -0.53] | -0.89 [-1.01 to -0.77] | -0.99 [-1.08 to -0.90]

ADVERSE EVENTS:
Time Frame: During the 2 week, double-blind treatment period, and up to and including 14 days (2 weeks) after the last dose of study therapy.
Description: Patients with two or more specific adverse experiences may be counted more than once in different categories, but only once in each category. Thus the count of Specific Other AEs may not add up to the count of Overall Other AEs.
Groups:
- Montelukast 10mg: Montelukast 10 mg tablet, loratadine matching-image placebo tablet, and montelukast/loratadine matching-image placebo tablet taken orally once daily at bedtime for 2 weeks.
- Loratadine 10mg: Montelukast matching-image placebo tablet, loratadine 10 mg tablet, and montelukast/loratadine matching-image placebo tablet taken orally once daily at bedtime for 2 weeks.
- Montelukast 10 mg + Loratadine 10 mg: Montelukast matching-image placebo tablet, loratadine matching-image placebo tablet, and montelukast 10 mg/loratadine 10 mg combination tablet taken orally once daily at bedtime for 2 weeks. During the study, patients in the montelukast/loratadine combination treatment group were discontinued from further participation due to a business decision by the sponsor.
Arm/Group | Placebo | Montelukast 10mg | Loratadine 10mg | Montelukast 10 mg + Loratadine 10 mg
Serious Adverse Events (participants affected / at risk) | 1/352 | 0/348 | 0/602 | 0/275
Other Adverse Events (participants affected / at risk) | 0/352 | 0/348 | 0/602 | 0/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=352) | Montelukast 10mg (N=348) | Loratadine 10mg (N=602) | Montelukast 10 mg + Loratadine 10 mg (N=275)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Montelukast/loratadine arm was discontinued due to business decision by sponsor to focus development on montelukast monotherapy. There was no efficacy data reported for this treatment arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.